CLINICAL TRIAL: NCT02614781
Title: Efficacy of Mifepristone - Prostaglandin Analogue Combination in Medical Termination of Pregnancy Beyond 7 Weeks of Amenorrhea
Status: Completed | Type: Observational
Sponsor: Nordic Pharma SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: RYMMA
Record Dates: First submitted 2015-11-20; First posted 2015-11-25 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Medical Termination of Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is a non-interventional prospective, multicenter, longitudinal study conducted in France, among a representative sample of public and/or private birth control centers.

The aim of the study is to assess, in real-life settings, the success rate of the protocol Mifegyne / prostaglandin analogue in patients asking for medical abortion either prior or beyond 7 weeks of amenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (≥ 18 years old) with confirmed intra-uterine pregnancy consulting for medical termination of pregnancy
* Patients for whom the physician decides to use a Mifegyne 600 mg and prostaglandin analogue combination for medical abortion
* Patients agreeing to participate in the study after having been informed orally by the physician and given the information sheet
* Informed patients accepting the computer processing of their medical data and their right of access and correction

Exclusion Criteria:

* Patients with known hypersensitivity to mifepristone
* Patients with known hypersensitivity to prostaglandin analogues (misoprostol or gemeprost).
* Patients with severe and progressive disease
* Patients with ectopic pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women asking for medical abortion
Sampling Method: Non-Probability Sample
Enrollment: 892 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
success rate of the protocol Mifegyne and prostaglandin analogue | At the follow-up at 2-3 weeks after inclusion
  The success rate will be defined as complete abortion without surgical procedure

SECONDARY OUTCOMES:
Success rate of the protocol Mifegyne and misoprostol per os. | at the follow up at 2-3 weeks after the inclusion
  The success rate will be defined as complete abortion without surgical procedure
rate of ongoing pregnancy by term. | at the follow up at 2-3 weeks after the inclusion
rate of patients requiring any additional procedures by term. | at the follow up at 2-3 weeks after the inclusion
Number of medical abortion using misoprostol | at the follow up at 2-3 weeks after the inclusion
  The number of medical abortion using misoprostol will be described.
Evaluation by patients of pain using a 5 level verbal rating scale | at the follow up at 2-3 weeks after the inclusion
  Physician will ask patients to evaluate the pain by a 5 level verbal rating scale. the using of pain killers will be also described

CONTACTS AND LOCATIONS:
Overall Officials: Hélène HERMAN-DEMARS, MD, Study Director — NORDIC PHARMA
Locations (1):
- Hôpital de la Conception, Marseille, France